CLINICAL TRIAL: NCT01538797
Title: YF476: Effects of a Single Dose at 3 Dose Levels on 24-hour Ambulatory Gastric pH Compared With Placebo and Ranitidine in Healthy Volunteers
Brief Title: Effect of Single Doses of YF476 on Stomach Acidity Compared With Ranitidine and Placebo in Fasted and Fed States
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 96-016
Record Dates: First submitted 2012-02-15; First posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Reflux Oesophagitis
Keywords: YF476; gastrin receptor antagonist; gastric pH; healthy subjects; ranitidine
MeSH Terms: conditions — Esophagitis, Peptic | interventions — YF 476; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YF476 — There were 5 treatments: 3 dose levels of YF476 (5, 25 and 100 mg), placebo and ranitidine 150 mg. There were at least 7 days between consecutive Treatment Days.
Drug: Ranitidine — There were 5 treatments: 3 dose levels of YF476 (5, 25 and 100mg), placebo and ranitidine 150mg. There were at least 7 days between consecutive Treatment Days.

SUMMARY:
The objectives of the study were:

* To compare a single dose of YF476 at 3 dose levels, placebo and ranitidine with respect to their effects on basal- and food- stimulated gastric pH in healthy volunteers.
* To assess whether there is a relationship between the pharmacokinetics of YF476 and gastric pH in healthy volunteers.
* To assess the safety and tolerability of single doses of YF476 in healthy volunteers.

DETAILED DESCRIPTION:
YF476 is clearly a potent and selective gastrin/CCK-B antagonist and should inhibit basal and meal-stimulated gastric acid secretion and enhance gastric emptying of a liquid meal in man. Therefore YF476 might benefit patients with reflux oesophagitis. The compound has been well tolerated in animal toxicity studies at doses in excess of the projected therapeutic dose in patients, and merits studies in healthy volunteers. Extrapolation from data obtained in animals suggests that a single oral dose of about 10mg of YF476 should compare favourably with an oral dose of 150mg of ranitidine in man with respect to effect on basal and food-stimulated gastric acid secretion. Therefore in the proposed study a range of doses of YF476 encompassing that dose will be studied; the exact dose of YF476 will be chosen on the basis of the previous study but the top dose will not exceed 100mg. 24-hour ambulatory gastric pH will be monitored via an intragastric pH electrode (7-10). Although there is variability between subjects with respect to the effects of food and drug treatment on gastric pH, the methodology for measurement of ambulatory gastric pH is robust.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and aged 18-45 years.
* No clinically relevant abnormal findings in the clinical history or physical examination at the screening assessment which could interfere with the objectives of the study or make the subject's participation hazardous.
* No clinically relevant abnormal laboratory values at the screening evaluation (Attachment 2).
* A normal ECG at the screening examination.
* A body mass index (Quetelet index) in the range 19-30:
* Body Mass Index = weight [kg]_ height [m]2
* Normal blood pressure and heart rate at the screening examination, i.e. BP 90-150mmHg systolic, 40-95mmHg diastolic; heart rate 40-100 beats/min in seated position.
* Subjects must be of sufficient intelligence to understand the nature of the study and any hazards of their participation in it. They must be able to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study.
* Subjects must give their written consent to participate after reading the Information-for-Volunteers Leaflet and Consent Form, and after having the opportunity to discuss the study with the Investigator or his deputy.

Exclusion Criteria:

* Females who are pregnant or lactating, or who are sexually active and are not using a reliable method of contraception.
* Clinically relevant abnormal history or physical findings at the screening assessment, which could interfere with the objectives of the study or the safety of the subject's participation.
* Clinically relevant abnormalities of laboratory values or ECG at screening evaluation.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate subject's participation in the study or make it unnecessarily hazardous.
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease or history of any psychotic mental illness.
* Participation in other clinical studies of a new chemical entity or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or intake of more than 40 units of alcohol weekly.
* Loss of more than 400mL blood during the 3 months before the study, e.g. as a blood donor.
* Use of prescription medication during 30 days before the study.
* Use of an over-the-counter medicine during 7 days before the study
* Blood pressure or heart rate outside those values specified under inclusion criterion (f).
* Possibility that the subject will not cooperate with the requirements of the protocol.
* Evidence of drug abuse on urine testing at study entry.
* Positive test for hepatitis B or C or HIV 1 & 2.
* High risk of hepatitis or HIV infection.
* History of severe allergic disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 1996-07; Primary Completion 1996-08 (Actual); Study Completion 1996-08 (Actual)

PRIMARY OUTCOMES:
Clinically relevant changes from baseline in safety assessments | 6 weeks
  Physical examination, ECG and safety tests of blood/urine at screening, 24h after dosing on each Treatment Day and at follow up. Blood pressure and heart rate before and at 0.5, 1, 2, 4, 6, 8, 12 and 24h after dosing on each Treatment Day.
Numbers of adverse events | 6 weeks
  Adverse events throughout the study
Pharmacokinetic parameters: Cmax, Tmax, AUC 0-24 h, T1/2 | 6 weeks
  Blood samples (8mL) before and at 0.5, 1, 2, 4, 6, 8, 12 and 24h after each dose for assay of YF476.
Pharmacodynamic parameters: continuous 24 h ambulatory gastric pH | 6 weeks
  Recording starts 0.5h before dosing on each Treatment Day; meals taken at 4, 9, 13 & 22h after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J Boyce, FRCP FFPM, Study Director — Trio Medicines Limited
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

REFERENCES:
- [Derived] Boyce M, David O, Darwin K, Mitchell T, Johnston A, Warrington S. Single oral doses of netazepide (YF476), a gastrin receptor antagonist, cause dose-dependent, sustained increases in gastric pH compared with placebo and ranitidine in healthy subjects. Aliment Pharmacol Ther. 2012 Jul;36(2):181-9. doi: 10.1111/j.1365-2036.2012.05143.x. Epub 2012 May 20. PMID 22607579